CLINICAL TRIAL: NCT04146350
Title: A Prospective Multicenter Study of Different Surgical Methods for the Treatment of Macular Schisis in High Myopia Based on the Real World
Brief Title: A Prospective Multicenter Study of Different Surgical Methods in the Treatment of High Myopic Macular Schisis
Acronym: Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AM1901D3
Record Dates: First submitted 2019-10-24; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Macular Schisis
MeSH Terms: interventions — Gases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (No Intervention)
- PPV+/-Cat (Active Comparator)
  Interventions: Procedure: PPV+/-Cat
- PPV+/-Cat+Gas (Active Comparator)
  Interventions: Procedure: PPV+/-Cat+Gas
- PPV+ILM+/-Cat+/-Gas (Active Comparator)
  Interventions: Procedure: PPV+ILM+/-Cat+/-Gas
- PPV+ILM+/-Cat+/-Oil (Active Comparator)
  Interventions: Procedure: PPV+ILM+/-Cat+/-Oil
- PSR (Active Comparator)
  Interventions: Procedure: PSR
- PSR+ PPV+ILM+/-Cat+/-Oil （or Gas） (Active Comparator)
  Interventions: Procedure: PSR+ PPV+ILM+/-Cat+/-Oil （or Gas）
- Gas (Active Comparator)
  Interventions: Procedure: Gas

INTERVENTIONS:
Procedure: PPV+/-Cat — pars plana vitrectomy+/-cataract
  Arms: PPV+/-Cat
Procedure: PPV+/-Cat+Gas — pars plana vitrectomy+/-cataract+gas tamponade
  Arms: PPV+/-Cat+Gas
Procedure: PPV+ILM+/-Cat+/-Gas — pars plana vitrectomy+internal limiting membrane peeling+/-cataract+/-gas tamponade
  Arms: PPV+ILM+/-Cat+/-Gas
Procedure: PPV+ILM+/-Cat+/-Oil — pars plana vitrectomy+internal limiting membrane peeling+/-cataract+/-silicone oil tamponade
  Arms: PPV+ILM+/-Cat+/-Oil
Procedure: PSR — posterior scleral reinforcement
  Arms: PSR
Procedure: PSR+ PPV+ILM+/-Cat+/-Oil （or Gas） — posterior scleral reinforcement+pars plana vitrectomy+internal limiting membrane peeling+/-cataract+/-silicone oil tamponade (or gas)
  Arms: PSR+ PPV+ILM+/-Cat+/-Oil （or Gas）
Procedure: Gas — gas tamponade alone
  Arms: Gas

SUMMARY:
In view of the current problem of treating high myopic macular schisis, the main purpose of our study is to find out the most appropriate time of surgical intervention, to compare the effectiveness and safety of various surgical methods in the treatment of high myopic macular schisis, and to find out the advantages and disadvantages of each surgical method in the treatment of MF. As well as the outcomes and complications of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. diopter ≤-6.00D or axial length ≥ 26.00mm;
2. OCT showed macular schisis with or without macular retinal detachment;
3. agreed to participate in this project and signed informed consent form.

Exclusion Criteria:

1. OCT confirmed full-thickness macular hole with or without macular retinal detachment；
2. submacular active or inactive CNV;
3. previous vitreoretinal surgery and anti-glaucoma surgery；
4. with rhegmatogenous retinal detachment, ocular trauma, glaucoma, corneal opacity and other ophthalmic diseases;
5. complicated with severe systemic disease can not tolerate surgery or follow-up;
6. do not agree to participate the project or disagree with the follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-10-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
foveal thickness | change from baseline foveal thickness at 3, 6, 9, 12 months
  measured by OCT
retinal thickness of the most significant schisis | change from baseline at 3, 6, 9, 12 months
  measured by OCT

SECONDARY OUTCOMES:
best corrected visual acuity | change from baseline at 3, 6, 9, 12 months
  BCVA
mf-ERG | change from baseline at 3, 6, 9, 12 months
  multifocal-ERG
Visual quality questionnaire | change from baseline at 3, 6, 9, 12 months
  Visual quality questionnaire
axial length | change from baseline at 3, 6, 9, 12 months
  axial length measured by IOL Master

CONTACTS AND LOCATIONS:
Overall Officials: Weisheng Li, Study Chair — Shanghai Aier Eye Hospital
Locations (1):
- Shanghai Aier Eye Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolar-Szczasny J, Swiech-Zubilewicz A, Mackiewicz J. A Review of Current Myopic Foveoschisis Management Strategies. Semin Ophthalmol. 2019;34(3):146-156. doi: 10.1080/08820538.2019.1610180. Epub 2019 May 6. PMID 31060414